CLINICAL TRIAL: NCT05204251
Title: Evaluation of the Quality of Life in Patients Referred for Transjugular Intrahepatic Portosystemic Shunt (TIPS) - Pilot Observational Cross-sectional Study
Brief Title: Evaluation of the Quality of Life in Patients Referred for Transjugular Intrahepatic Portosystemic Shunt
Acronym: TIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8338
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Liver Disease
Keywords: Chronic liver disease; TIPS; Quality of life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — Quality of Life assessed with the SF-36 questionnaire

SUMMARY:
Patient with Advanced Chronic Liver Disease often present portal hypertension which may lead to bleading or ascites.

One of the treatment of portal hypertension in these patients is the placement of a Transjugular Intrahepatic Portosystemic Shunt (TIPS).

The indications for placing TIPS take on various clinical presentations, the most classic being digestive haemorrhage by rupture of oesophageal and/or gastric varices and refractory ascites.

TIPS placement involves changes in haemodynamics and liver function that may alter the patients' condition and quality of life.

Very few articles have evaluated the quality of life of these patients and when quality of life is evaluated it is mostly with not adapted or not validated scales.

The main objective of this study is to evaluate the quality of life of patients who have undergone TIPS using a validated and standardised quality of life questionnaire (the SF-36 questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients referred to the TIPS service between January 2012 and October 2020 at the University Hospitals of Strasbourg, with a follow-up period of at least 1 month
* Subjects who have not expressed any opposition to the use of their medical data for research purposes
* For subjects invited to fill in the questionnaires: subject having expressed his/her agreement with the use of his/her medical data in the framework of the current study

Exclusion Criteria:

* Diseased patient
* Liver transplant patient following TIPS
* Pregnancy
* Patient in a vulnerable situation
* Patient under court protection, guardianship or trusteeship
* Difficulties in understanding the questionnaire
* Impossible to give the subject informed information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Advanced Chronic Liver Disease who underwent a Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement at the University Hospital of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Mental component of quality of Life of the | 45 minutes
  Assessment of the mental component of quality of life by a generic questionnaire (SF-36),

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie Interventionnelle Vasculaire - CHU de Strasbourg - France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided